CLINICAL TRIAL: NCT06263361
Title: Improving Safety and Accuracy of Stereotactic Brain Biopsies in Primary Central Nervous System Lymphoma (PCNSL): Integration of Advanced MRI Patterns and Fluorescein Sodium Fluorescence
Brief Title: Improving Safety and Accuracy of Stereotactic Brain Biopsies in Primary Central Nervous System Lymphoma.
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Pietro Mortini, MD, Prof., Professor, Head of Department, IRCCS San Raffaele
Other Study IDs: NCH02-2021
Record Dates: First submitted 2024-01-30; First posted 2024-02-16 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Included patients: Adult patients (>18 years) candidates to stereotactic biopsy for histopathological diagnosis of intra-axial lesions suspected for primary central nervous system lymphoma (PCNSLs).
  Interventions: Diagnostic Test: MRI imaging; Diagnostic Test: Cerebral biopsy

INTERVENTIONS:
Diagnostic Test: MRI imaging — To characterize the peritumoral area in PCNLs through the use of advanced MRI sequences.
Diagnostic Test: Cerebral biopsy — To evaluate the predictive value of sodium fluorescence to confirm ex-vivo the diagnostic tumor tissue prior to histopathological examination.

SUMMARY:
Primary central nervous system lymphoma (PCNSL) is an aggressive extranodal non- Hodgkin lymphoma exclusively localized into the nervous system. The aim of this study is to evaluate the MRI imaging characteristics of the peritumoral area (PTA) and to correlate this information to pathological findings.

DETAILED DESCRIPTION:
Primary central nervous system lymphoma (PCNSL) is an aggressive extranodal non- Hodgkin lymphoma exclusively localized into the nervous system. It is a relatively rare disorder, accounting for only 3% of all primary brain tumors but due to its anatomical localization represents an important clinical and diagnostic challenge in onco-hematology. different MRI patterns of the peritumoral area (PTA) might correlate with different histopathological sensitivity regarding diagnostic potential out of contrast-enhanced region (CER). Improvements in the understanding of PTA diagnostic potentials is of great help in diagnosing patients with deep-seated lesions, who would otherwise be not eligible for stereotactic biopsy and therefore for a consequent adequate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, undergoing stereotactic biopsy for newly diagnosed PSNCLs

Exclusion Criteria:

* Severe hepatic dysfunction
* Severe renal dysfunction
* Severe heart failure
* myocardial infarction and stroke within 90 days
* Hyperreactivity against contrast agents
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, undergoing stereotactic biopsy for newly diagnosed PSNCLs at our Institution, able to express informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI imaging | Baseline (before surgery)
  Peritumoral area (PTA) volumes in T1w sequence Units: cm3.
MRI imaging | Baseline (before surgery)
  Peritumoral area (PTA) volumes in T2w sequence. Units: cm3.
MRI imaging | Baseline (before surgery)
  Peritumoral area (PTA) volumes in FLAIR sequence. Units: cm3.
MRI imaging | Baseline (before surgery)
  Peritumoral area (PTA) mean ADC value in PTA. Units: mm2/s
Define immunopathological features | 1 week after surgical procedure
  Number of immune cells infiltrating the lesion. Units: number/mm3

SECONDARY OUTCOMES:
Accuracy of fluoresceine guided stereotactic biopsy | 1 week after surgical procedure
  Number of patients with samples positively stained with fluoresceine. Units: number of samples/patients

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Mortini, MD, Prof., Study Director — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akshulakov SK, Kerimbayev TT, Biryuchkov MY, Urunbayev YA, Farhadi DS, Byvaltsev VA. Current Trends for Improving Safety of Stereotactic Brain Biopsies: Advanced Optical Methods for Vessel Avoidance and Tumor Detection. Front Oncol. 2019 Oct 2;9:947. doi: 10.3389/fonc.2019.00947. eCollection 2019. PMID 31632903
- [Background] Barajas RF Jr, Rubenstein JL, Chang JS, Hwang J, Cha S. Diffusion-weighted MR imaging derived apparent diffusion coefficient is predictive of clinical outcome in primary central nervous system lymphoma. AJNR Am J Neuroradiol. 2010 Jan;31(1):60-6. doi: 10.3174/ajnr.A1750. Epub 2009 Sep 3. PMID 19729544
- [Background] Barajas RF, Politi LS, Anzalone N, Schoder H, Fox CP, Boxerman JL, Kaufmann TJ, Quarles CC, Ellingson BM, Auer D, Andronesi OC, Ferreri AJM, Mrugala MM, Grommes C, Neuwelt EA, Ambady P, Rubenstein JL, Illerhaus G, Nagane M, Batchelor TT, Hu LS. Consensus recommendations for MRI and PET imaging of primary central nervous system lymphoma: guideline statement from the International Primary CNS Lymphoma Collaborative Group (IPCG). Neuro Oncol. 2021 Jul 1;23(7):1056-1071. doi: 10.1093/neuonc/noab020. PMID 33560416
- [Background] Harris N, Fetter RD, Brasier DJ, Tong A, Davis GW. Molecular Interface of Neuronal Innate Immunity, Synaptic Vesicle Stabilization, and Presynaptic Homeostatic Plasticity. Neuron. 2018 Dec 5;100(5):1163-1179.e4. doi: 10.1016/j.neuron.2018.09.048. Epub 2018 Oct 18. PMID 30344041
- [Background] Chen B, Wang H, Ge P, Zhao J, Li W, Gu H, Wang G, Luo Y, Chen D. Gross total resection of glioma with the intraoperative fluorescence-guidance of fluorescein sodium. Int J Med Sci. 2012;9(8):708-14. doi: 10.7150/ijms.4843. Epub 2012 Oct 6. PMID 23091408
- [Background] Acerbi F, Broggi M, Schebesch KM, Hohne J, Cavallo C, De Laurentis C, Eoli M, Anghileri E, Servida M, Boffano C, Pollo B, Schiariti M, Visintini S, Montomoli C, Bosio L, La Corte E, Broggi G, Brawanski A, Ferroli P. Fluorescein-Guided Surgery for Resection of High-Grade Gliomas: A Multicentric Prospective Phase II Study (FLUOGLIO). Clin Cancer Res. 2018 Jan 1;24(1):52-61. doi: 10.1158/1078-0432.CCR-17-1184. Epub 2017 Oct 10. PMID 29018053
- [Background] Hamamcioglu MK, Akcakaya MO, Goker B, Kasimcan MO, Kiris T. The use of the YELLOW 560 nm surgical microscope filter for sodium fluorescein-guided resection of brain tumors: Our preliminary results in a series of 28 patients. Clin Neurol Neurosurg. 2016 Apr;143:39-45. doi: 10.1016/j.clineuro.2016.02.006. Epub 2016 Feb 11. PMID 26895208
- [Background] Koc K, Anik I, Cabuk B, Ceylan S. Fluorescein sodium-guided surgery in glioblastoma multiforme: a prospective evaluation. Br J Neurosurg. 2008 Feb;22(1):99-103. doi: 10.1080/02688690701765524. PMID 18224529
- [Background] Li Y, Rey-Dios R, Roberts DW, Valdes PA, Cohen-Gadol AA. Intraoperative fluorescence-guided resection of high-grade gliomas: a comparison of the present techniques and evolution of future strategies. World Neurosurg. 2014 Jul-Aug;82(1-2):175-85. doi: 10.1016/j.wneu.2013.06.014. Epub 2013 Jul 9. PMID 23851210